CLINICAL TRIAL: NCT00525668
Title: Sunphenon EGCg (Epigallocatechin-gallate) in Relapsing-remitting Multiple Sclerosis (SuniMS Study)
Brief Title: Sunphenon Epigallocatechin-gallate (EGCg) in Relapsing-remitting Multiple Sclerosis (SuniMS Study)
Acronym: SuniMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Friedemann Paul, Prof., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-006323-39
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: multiple sclerosis; inflammation; neurodegeneration; neuroprotection
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Inflammation; Nerve Degeneration | interventions — epigallocatechin gallate; Sunphenon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- verum (Active Comparator): Sunphenon plus glatiramer acetate
  Interventions: Drug: epigallocatechin-gallate (Sunphenon)
- placebo (Active Comparator): placebo plus glatiramer acetate
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: epigallocatechin-gallate (Sunphenon) — 200 mg twice daily, after 3 months 400 mg twice daily
  Arms: verum
Drug: placebo — 2 placebo capsules twice daily, after 3 months 4 placebo capsules twice daily
  Arms: placebo

SUMMARY:
Hypothesis:

Sunphenon, a green tea extract containing 95% egcg, given daily as oral medication over a period of 18 months has anti-inflammatory and neuroprotective properties in patients with relapsing-remitting multiple sclerosis as assessed by magnetic resonance imaging and clinical examination (EDSS and MSFC).

DETAILED DESCRIPTION:
This multicentric, national study investigates the efficacy and safety of EGCG in patients with relapsing-remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects age 18 to 60
* relapsing-remitting course of MS
* stable treatment with glatiramer acetate at least 6 months prior to inclusion

Exclusion Criteria:

* primary or secondary progressive forms of MS
* clinically relevant heart, lung, liver, kidney diseases
* regular hepatotoxic co-medication
* drug addiction
* alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
number of new T2 lesions on brain MRI performed after 18 months of Sunphenon treatment compared to baseline MRI in the verum arm versus placebo | 18 months

SECONDARY OUTCOMES:
development of brain atrophy under treatment with EGCG vs. placebo | 18 months
Safety and tolerability | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Bellmann-Strobl, Dr., MD, Principal Investigator — Experimental and Clinical Research Center, Charite University, Berlin, Germany; Friedemann Paul, Prof., MD, Study Director — NeuroCure Clinical Research Center, Charité University, Berlin, Germany
Locations (2):
- Germany (2):
  - NeuroCure Clinical Research Center, Charite University, Berlin, Berlin
  - Outpatient Clinic for Neuroimmunology at the ECRC, Charite University, Berlin, Berlin

REFERENCES:
- [Derived] Bellmann-Strobl J, Paul F, Wuerfel J, Dorr J, Infante-Duarte C, Heidrich E, Kortgen B, Brandt A, Pfuller C, Radbruch H, Rust R, Siffrin V, Aktas O, Heesen C, Faiss J, Hoffmann F, Lorenz M, Zimmermann B, Groppa S, Wernecke KD, Zipp F. Epigallocatechin Gallate in Relapsing-Remitting Multiple Sclerosis: A Randomized, Placebo-Controlled Trial. Neurol Neuroimmunol Neuroinflamm. 2021 Mar 24;8(3):e981. doi: 10.1212/NXI.0000000000000981. Print 2021 May. PMID 33762428
- See also: Homepage of the NeuroCure Clinical Research Center — http://www.ncrc.de